CLINICAL TRIAL: NCT02495844
Title: Double-blind, Randomized, Placebo-controlled Study of the Efficacy, Safety/Tolerability, and Pharmacokinetic Profile of UCB0942 in Adults With Highly Drug-resistant Focal Epilepsy.
Brief Title: A Study of UCB0942 in Adult Patients With Highly Drug-resistant Focal Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP0069; 2014-003330-12 (EudraCT Number)
Record Dates: First submitted 2015-06-29; First posted 2015-07-13 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Highly Drug-resistant Focal Epilepsy
Keywords: UCB0942; Treatment-resistant focal epilepsy; Partial seizures; Seizure therapy
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UCB0942 (Experimental): UCB0942/UCB0942
  Interventions: Drug: UCB0942
- Placebo (Placebo Comparator): Placebo/UCB0942 (after 2-week inpatient period, placebo subjects will receive the experimental medicine, UCB0942).
  Interventions: Drug: UCB0942; Drug: Placebo

INTERVENTIONS:
Drug: UCB0942 — Active substance: UCB0942 Pharmaceutical form: Film-coated tablet Concentration: 200 mg Route of Administration: Oral use
  Arms: UCB0942
Drug: UCB0942 — Active substance: UCB0942 Pharmaceutical form: Film-coated tablet Concentration: 100 mg Route of Administration: Oral use
Drug: Placebo — Pharmaceutical form: Film-coated tablet Route of administration: Oral use
  Arms: Placebo

SUMMARY:
This study is to assess the efficacy, safety, and tolerability of the investigational drug UCB0942in adult subjects with drug-resistant focal epilepsy across multiple centers in Europe.

DETAILED DESCRIPTION:
The study will include a Screening Visit, a Prospective Outpatient Baseline Period (2 to 3 weeks), an Inpatient Period (3 weeks), an Outpatient Period (8 weeks of treatment and 2 weeks of taper), and a Safety Follow-Up Period (4 weeks). The total study duration after screening will be 19 to 20 weeks. Approximately 6 months after the last visit subjects will be asked to return for an additional visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult (18 years of age or more)
* Subject is able to understand the study and the ICF as assessed by the Investigator. Subjects with known mental retardation (defined as IQ below 70) are not eligible to participate. Subject and/or caregiver is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, and the medication intake scheme as instructed according to the judgment of the Investigator
* Subject fulfills ILAE (1989) criteria for focal epilepsy; clinical semiology should be described and fulfill criteria for focal seizures; there will have been an electroencephalogram (EEG) reading compatible with focal epilepsy in the last 5 years; the subject has no seizures that are not focal by the new ILAE criteria; a brain MRI (magnetic resonance imaging) or head CT (computed tomography) to be performed before randomization, if no such scan was performed in the last 5 years, and a report is available. If a scan was performed within the last 5 years but the epilepsy has not been stable since the last scan, a new scan should be obtained
* Subject has failed to achieve seizure control with ≥4 appropriately chosen Antiepileptic Drug (AED) regimens of adequate dose and duration, including the current treatment, as documented in medical records and per Investigator assessment of patient report
* Subject is currently treated with a stable dose of at least 1 AED for the 4 weeks prior to the Screening Visit (Visit 1) and throughout the duration of the Treatment Period with or without additional concurrent vagus nerve stimulation (VNS) or other neurostimulation treatments. The VNS must have been in place for at least 12 months with constant settings for at least 3 months and the battery life of unit anticipated to extend for the duration of study prior to the Screening Visit and throughout the duration of the study
* During the 4 weeks prior to Screening (Historical Baseline Period), subject must report to have had an average of at least 4 spontaneous and observable focal seizures per week ("focal seizures" refers to partial-onset seizures of type IA1, IB, and IC, but does not include type IA2, IA3, or IA4 seizures), and cannot have had any seizure-free period longer than 3 days (based on Investigator assessment of subject report and seizure diaries if available). The cut-off seizure frequency (4 seizures per week) and maximum seizure-free interval (3 days) must be maintained during the 2-week Prospective Outpatient Baseline Period
* Female subjects of nonchildbearing potential (premenarcheal, postmenopausal for at least 2 years, bilateral oophorectomy or tubal ligation, and complete hysterectomy) are eligible. Female subjects of childbearing potential are eligible if they use medically accepted contraceptive methods. Oral or depot contraceptive treatment with at least ethinylestradiol 30 μg per intake used with an additional barrier contraception method, monogamous relationship with vasectomized or female partner, or double-barrier contraception are acceptable methods. The subject must understand the consequences and potential risks of inadequately protected sexual activity, be educated about and understand the proper use of contraceptive methods, and undertake to inform the Investigator of any potential change in status. Abstinence will be considered as an acceptable method of contraception if the Investigator can document that the subject agrees to be compliant when it is in line with the preferred and usual lifestyle of the subject
* Male subjects confirm that during the study period and for a period of 3 months after the final dose, when having sexual intercourse with a woman of childbearing potential, he will use a barrier contraceptive (eg, condom) and that the respective partner will use an additional contraceptive method

Exclusion Criteria:

* Subject has participated in another study of an investigational medication (or medical device) within the last 30 days or is currently participating in another study of an investigational medication (or a medical device)
* Subject has a known hypersensitivity to any components of UCB0942 formulation or to similar drugs (LEV, BRV, or benzodiazepines), or a history of drug or other allergy that, in the opinion of the Investigator or UCB Study Physician, contraindicates her/his participation
* Subject has a current or past psychiatric condition that, in the opinion of the Investigator, could compromise his/her safety or ability to participate in this study including a history of schizophrenia, schizoaffective disorder, bipolar disorder, or severe unipolar depression. The presence of potential psychiatric exclusion criteria will be determined based on screening with the BPRS plus the Mini International Neuropsychiatric Interview (MINI)
* Subject has taken other (non-AED) prescription, nonprescription, dietary (eg, grapefruit or passion fruit), or herbal products that are potent inducers or inhibitors of the CYP3A4 pathway for 2 weeks (or 5 half-lives, whichever is longer) prior to the Baseline Visit
* Subject is currently treated with carbamazepine, phenytoin, primidone, or phenobarbital or any other drug known to induce CYP3A4 liver enzymes; Subject is taking tiagabine, felbamate, or vigabatrin; Subject is taking benzodiazepines, zolpidem, zaleplon, or zopiclone >3 times per week for any indication
* Subject has a clinically significant abnormality on echocardiography at Screening or a history of rheumatic heart disease or other known valvular abnormalities
* Subjects with a history of hypersensitivity reactions or autoimmune disease
* Female subject who is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (18):
- Belgium (3):
  - Ep0069 103, Brussels
  - Ep0069 101, Ghent
  - Ep0069 102, Leuven
- Ep0069 201, Sofia, Bulgaria
- Germany (6):
  - Ep0069 402, Bielefeld
  - Ep0069 408, Hamburg
  - Ep0069 401, Kehlkork
  - Ep0069 407, Marburg
  - Ep0069 403, Radeberg
  - Ep0069 405, Ravensburg
- Hungary (2):
  - Ep0069 601, Budapest
  - Ep0069 602, Budapest
- Ep0069 302, Heeze, Netherlands
- Spain (5):
  - Ep0069 502, Barcelona
  - Ep0069 505, Llobregat
  - Ep0069 506, Madrid
  - Ep0069 501, Seville
  - Ep0069 503, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in August 2015 and concluded in July 2017.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Groups:
- Placebo/UCB0942: After 2-week in the Inpatient Period, Placebo subjects received the experimental medicine (UCB0942).
- UCB0942/UCB0942: Subjects received UCB0942.
Period: Overall Study
Arm/Group | Placebo/UCB0942 | UCB0942/UCB0942
Started | 27 | 28
Completed | 26 | 24
Not Completed | 1 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — AE, non-fatal | 0 | 1
Not completed — Hepatitis Positivity | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set consisting of all subjects in the Randomized Set who received at least 1 dose of Investigational Medicinal Product (IMP).
Arm/Group | Placebo/UCB0942 | UCB0942/UCB0942 | Total Title
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (8.7) | 36.2 (11.4) | 35.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 27 | 25 | 52
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 26 | 25 | 51
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.66 (4.82) | 27.20 (4.32) | 26.45 (4.59)

OUTCOME MEASURES:

1. Primary Outcome: 75 % Responder Rate During the 2-week Inpatient Period
Description: The 75% responder rate is defined as the percentage of subjects with a 75 % or greater reduction in focal seizure frequency during the 2-week Inpatient Period compared with the Baseline Period.
Time Frame: During the 2-week Inpatient Period
Measure: Number; unit: percentage of participants
Groups:
- Placebo/UCB0942 (FAS): After 2-week in the Inpatient Period, Placebo subjects received the experimental medicine (UCB0942).
- UCB0942/UCB0942 (FAS): Subjects received UCB0942.
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 26
percentage of participants | 11.1 | 30.8
Statistical Analysis 1: Comparison: Placebo/UCB0942 (FAS) vs UCB0942/UCB0942 (FAS); Test type: Superiority; p = 0.0679, Regression, Logistic; Odds Ratio (OR) = 4.14, 95% CI 2-sided [0.90 to 19.06]

2. Secondary Outcome: Median Percent Change in Weekly Focal Seizure Frequency During the 2-week Inpatient Period
Description: A negative value in median percent change reflects a reduction from Baseline.
Time Frame: During the 2-week Inpatient Period
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 26
percentage of change | -12.5 [-57.14 to 41.11] | -53.68 [-84.61 to -22.73]

3. Secondary Outcome: Median Percent Change in Weekly Focal Seizure Frequency During the Outpatient Maintenance Period
Description: A negative value in median percent change reflects a reduction from Baseline.
Time Frame: During the Outpatient Maintenance Period (8 weeks)
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 25
percentage of change | -57.94 [-76.23 to -29.09] | -26.32 [-77.38 to -3.07]

4. Secondary Outcome: Median Percent Change in Weekly Focal Seizure Frequency During the On-UCB0942 Overall Period
Description: A negative value in median percent change reflects a reduction from Baseline.
Time Frame: During the On-UCB0942 Overall Period (approximately 11 weeks)
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 27
percentage of change | -53.85 [-78.01 to -34.48] | -29.87 [-76.39 to -11.36]

5. Secondary Outcome: Seizure-free Rate (All Seizures) During the 2-week Inpatient Period
Description: Seizure-free rate is reported as the percentage of seizure-free participants during the 2-week Inpatient Period.
Time Frame: During the 2-week Inpatient Period
Measure: Number; unit: percentage of particpants
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 27
percentage of particpants | 3.7 | 7.4

6. Secondary Outcome: Seizure-free Rate (All Seizures) During the Last 4 Weeks of the Outpatient Maintenance Period
Description: Seizure-free rate is reported as the percentage of seizure-free participants during the last 4 weeks of the Outpatient Maintenance Period.
Time Frame: During the last 4 weeks of the Outpatient Maintenance Period
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 25
percentage of participants | 0 | 0

7. Secondary Outcome: Seizure-free Rate (All Seizures) During the On-UCB0942 Overall Period
Description: Seizure-free rate is reported as the percentage of seizure-free participants during the On-UCB0942 Overall Period.
Time Frame: During the On-UCB0942 Overall Period (approximately 11 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 28
percentage of participants | 0 | 0

8. Secondary Outcome: 75 % Responder Rate During the Last 4 Weeks of the Outpatient Maintenance Period
Description: The 75 % responder rate is defined as the percentage of subjects who achieve a 75 % or greater reduction in focal seizure frequency.
Time Frame: During the last 4 weeks of the Outpatient Maintenance Period
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 24
percentage of participants | 33.3 | 29.2

9. Secondary Outcome: 75 % Responder Rate During the On-UCB0942 Overall Period
Description: as for outcome 8
Time Frame: During the On-UCB0942 Overall Period (approximately 11 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 27
percentage of participants | 25.9 | 25.9

10. Secondary Outcome: Percentage of Seizure Free Days (All Seizures) During the 2-week Inpatient Period
Description: For the active group, the 2-week Inpatient Period refers to the last 2 weeks of the Inpatient Period, while for the Placebo group, it refers to the first 2 weeks of the Inpatient Period.
Time Frame: During the 2-week Inpatient Period
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 27
percentage of days | 21.43 [7.14 to 57.14] | 57.14 [28.57 to 78.57]

11. Secondary Outcome: Percentage of Seizure-free Days (All Seizures) During the Outpatient Maintenance Period
Time Frame: During the Outpatient Maintenance Period (8 weeks)
Measure: Median (Inter-Quartile Range); unit: percentage of days
Arm/Group | Placebo/UCB0942 (FAS) | UCB0942/UCB0942 (FAS)
Number analyzed (Participants) | 27 | 26
percentage of days | 51.79 [15.79 to 80.70] | 51.35 [29.82 to 69.64]

12. Secondary Outcome: Number of Patients Reporting at Least One Serious Adverse Event (SAE) During the Course of the Study
Description: Number of subjects experiencing at least one serious adverse event (reported by the subject and/or caregiver or observed by the Investigator or inpatient staff).
Time Frame: All study duration (approximately 19 to 20 weeks)
Measure: Number; unit: Participants
Groups:
- Placebo/UCB0942 (SS): After 2-week in the Inpatient Period, Placebo subjects received the experimental medicine (UCB0942).
- UCB0942/UCB0942 (SS): Subjects received UCB0942.
Arm/Group | Placebo/UCB0942 (SS) | UCB0942/UCB0942 (SS)
Number analyzed (Participants) | 27 | 28
Participants | 0 | 2

13. Secondary Outcome: Number of Subject Withdrawals Due to Adverse Events (AEs) During the Course of the Study
Description: Number of subjects who withdrew from the study due adverse event (reported by the subject and/or caregiver or observed by the Investigator or inpatient staff).
Time Frame: All study duration (approximately 19 to 20 weeks)
Measure: Number; unit: Participants
Arm/Group | Placebo/UCB0942 (SS) | UCB0942/UCB0942 (SS)
Number analyzed (Participants) | 27 | 28
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Baseline until Safety Follow Up Visit (up to Week 28).
Description: Baseline Characteristics refer to the Safety Set consisting of all subjects in the Randomized Set who received at least 1 dose of Investigational Medicinal Product (IMP). 2 subjects reported multiple Serious Adverse Events (SAEs).
Arm/Group | Placebo/UCB0942 | UCB0942/UCB0942
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/28
Other Adverse Events (participants affected / at risk) | 26/27 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/UCB0942 (N=27) | UCB0942/UCB0942 (N=28)
Judgement impaired (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/UCB0942 (N=27) | UCB0942/UCB0942 (N=28)
Somnolence (Nervous system disorders) | 12 (16) | 17 (24)
Dizziness (Nervous system disorders) | 12 (51) | 14 (19)
Headache (Nervous system disorders) | 6 (9) | 10 (13)
Tremor (Nervous system disorders) | 3 (3) | 2 (2)
Disturbance in attention (Nervous system disorders) | 1 (2) | 3 (3)
Dysarthria (Nervous system disorders) | 2 (2) | 3 (5)
Memory impairment (Nervous system disorders) | 1 (2) | 3 (6)
Nystagmus (Nervous system disorders) | 3 (3) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (2) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 3 (3)
Simple partial seizures (Nervous system disorders) | 1 (1) | 2 (5)
Ataxia (Nervous system disorders) | 0 (0) | 2 (3)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 4 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (5)
Depressed mood (Psychiatric disorders) | 1 (1) | 2 (2)
Nervousness (Psychiatric disorders) | 2 (3) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 2 (3)
Mood swings (Psychiatric disorders) | 0 (0) | 2 (2)
Parasomnia (Psychiatric disorders) | 0 (0) | 2 (3)
Aggression (Psychiatric disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 9 (14) | 4 (23)
Gait disturbance (General disorders) | 2 (2) | 3 (17)
Asthenia (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 2 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Muscosloskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 3 (4)
Hypotension (Vascular disorders) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT02495844/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT02495844/SAP_001.pdf